CLINICAL TRIAL: NCT03398460
Title: Burnout and Approach to Bereavement Initiatives in a Medical Intensive Care Unit (ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-01695
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional | interventions — Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Care Providers (Other): Bellevue hospital Medical Intensive Care Unit; 30 Nurses and 50 physcians
  Interventions: Diagnostic Test: Survey

INTERVENTIONS:
Diagnostic Test: Survey — Burnout rates before and after the introduction of a bereavement card Burnout rates before and after an ICU rotation for physicians

SUMMARY:
Given the stress, exhaustion and close interface with death that Intensive Care Unit (ICU) health care providers face, this study will evaluate burnout rates in intensive care unit (icu) physicians, nurses and ancillary staff. Investigators will also study the effect on a bereavement card on these burnout rates

DETAILED DESCRIPTION:
This study will evaluate:

1. Burnout rates among nurses and ancillary staff with the Abbreviated Maslach burnout inventory. This is a well validated tool that is used to evaluate symptoms of burnout such as denationalization, emotional exhaustion and lack of personal accomplishment.
2. Burnout rates at the beginning of and at the end of the house staff's ICU rotation to gauge the effect of an ICU rotation on burnout rates amon medical trainees.
3. Determine whether the introduction of a bereavement card will improve symptoms of burnout as gauged by the abbreviated maslach burnout inventory
4. Staff perceptions and response to the introduction of a bereavement

ELIGIBILITY:
Inclusion Criteria:

* Health care providers who work in the Bellevue Hospital Medical ICU

Exclusion Criteria:

* NA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Burnout rate before introduction of bereavement card | 1 Year
  Measured by "Staff Response Questionnaire"
Burnout rate after introduction after introduction of bereavement card | 1 Year
  Measured by "Staff Response Questionnaire"
Burnout rates before ICU rotation for physicians | 1 Year
  Measured by "Staff Response Questionnaire"
Burnout rates after an ICU rotation for physicians | 1 Year
  Measured by "Staff Response Questionnaire"

CONTACTS AND LOCATIONS:
Overall Officials: Vikramjit Mukherjee, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States